CLINICAL TRIAL: NCT04767074
Title: A Non-pharmacological Cough Control Therapy as an Adjuvant of Pulmonary Rehabilitation in People With Interstitial Lung Diseases and Chronic Cough - A Feasibility Study
Brief Title: A Non-pharmacological Cough Control Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Dina Brooks, Senior Scientist, West Park Healthcare Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-005-WP
Record Dates: First submitted 2021-02-18; First posted 2021-02-23 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Cough; ILD; Pulmonary Disease; Pulmonary Fibrosis
Keywords: Cough; ILD; Pulmonary rehabilitation; chronic cough; non-pharmacological cough therapy
MeSH Terms: conditions — Cough; Lung Diseases; Pulmonary Fibrosis; Chronic Cough

STUDY DESIGN:
Intervention Model Description: Feasibility Pre/Post interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-pharmacological Cough control therapy (Experimental): Participants will attend four virtual sessions of 45 to 60 minutes of educational and self-management. Sessions will be designed to target participants' needs and expectations according to the semi-structured theme.
  Session 1 General assessment Prescription of cough technique
  Session 2 Cough principles of cough Cough control
  Session 3 Breathing pattern retraining and laryngeal hygiene
  Session 4 Reinforcement of cough control therapies
  Interventions: Other: Non-pharmacological Cough control Therapy

INTERVENTIONS:
Other: Non-pharmacological Cough control Therapy — Participants will attend four virtual sessions of 45 to 60 minutes of educational and self-management.
  Session 1 General assessment Prescription and taught of one cough suppression technique.
  Session 2 Cough principles: mechanism, cough reflex, chronic cough, the importance of cough and negative effects of repeated coughing.
  Cough control: identify triggers, use cough suppressions and distractions techniques.
  Session 3 Breathing pattern retraining and laryngeal hygiene: reinforce nasal breathing and pursed lips breathing as strategies to avoid the urge to cough, identification of risk factors for laryngeal dehydration and hydration education.
  Session 4 Reinforcement: Clarification of doubts, techniques' reinforcement and application during daily life situations.
  Other Names: Cough Control therapy

SUMMARY:
Coughing affects almost all individuals with ILD leading to physical, psychological and social distress and prevents individuals from performing their activities of daily living, working or socialising in public places. Unfortunately, there are no licensed medications available to treat chronic cough and the few drugs that have been tried resulted in little efficacy and significant side effects. Drug-free cough control interventions have shown promise in reducing the severity and impact of coughing on patients' lives but have not been tested in individuals with ILD. This study aims to explore the feasibility and effectiveness of a non-pharmacological cough control therapy, as an adjuvant of pulmonary rehabilitation, in patients with ILD and chronic cough (>8 weeks in duration).

DETAILED DESCRIPTION:
Research questions and hypotheses

i) Is a non-pharmacological cough control therapy feasible to treat chronic cough in patients with ILD? Hypothesis: Given the results of previous non-pharmacological interventions in patients with refractory cough, we predict that this intervention will be feasible and well accepted in patients with ILD.

ii) Is a non-pharmacological cough control therapy more effective than pulmonary rehabilitation (PR) alone to treat chronic cough in patients with ILD? Hypotheses: Given the results of previous non-pharmacological interventions in patients with refractory cough, we predict that improvements observed in participants receiving the non-pharmacological intervention will exceed those receiving PR alone. Improvements are expected in HRQOL (exceeding the minimal clinically important difference), intensity of cough-related sensations and symptoms of fatigue.

Research Design The proposed research is a feasibility pre-post intervention study.

Study details:

Adults with ILD and chronic cough will be enrolled in this study. Potential eligible patients will be recruited from the outpatient PR program at West Park Healthcare Centre and St. Joseph's Healthcare. As the outpatient pulmonary rehabilitation program at West Park Healthcare Center and St. Joseph's Healthcare will transition partially to virtual meetings, the interactions between the research team and patients will be completed via phone calls or online.

This research study will be delivered online using the Zoom Healthcare Plan, an online platform that is available at West Park Healthcare Centre, and is used for telerehabilitation programs. Participants will be enrolled into a PR program composed of aerobic and strengthening exercises, disease-specific education and self-management, as part of their usual care. Two weeks before termination of PR, participants will start the non-pharmacological cough control therapy, following the intervention proposed by Chamberlain colleagues (2017). Participants will attend four virtual sessions of 45 to 60 minutes of educational and self-management

This study will measure several clinical outcomes.

1. Feasibility will be reflected by the number of eligible patients enrolling (enrolment rate of at least 75%) and completing the intervention (attendance rate of at least 80%), compliance with the sessions and adverse events.
2. Leicester cough questionnaire
3. The King's Brief Interstitial Lung Disease (KBILD)
4. Modified Borg scale (mBorg
5. Cough Hypersensitivity Questionnaire (CHQ)
6. Functional Assessment of Chronic Illness Therapy Fatigue Scale (FACIT-F)
7. Global rating of change questionnaire (GRCQ)
8. Satisfaction Semi-structured interviews using open-ended questions will be conducted before and after the cough control intervention to capture participants' expectations and perspectives about the cough control therapy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals will be included if having confirmed diagnosis of any ILD by a physician (as per Canadian Thoracic Society's guideline for evaluating patients with fibrotic interstitial lung disease) and a chronic cough lasting more than 8 weeks in duration

Exclusion Criteria:

* self-reports of moderate or large sputum production
* effective or suspected exacerbation of the respiratory condition in the past month
* upper respiratory tract infection in the past month
* use of angiotensin-converting enzyme inhibitor medication
* changes in the prescribed medication in the previous month
* evidence of traction bronchiectasis in the HRCT
* evidence of other medical conditions that prevent performance of an exercise training program
* unable to read or speak in English / unable to provide informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intervention | through study completion, average 1 year
  intervention feasibility will be reflected by the number of eligible patients enrolling (enrolment rate of at least 75%) and completing the intervention (attendance rate of at least 80%), compliance with the sessions and adverse events.

SECONDARY OUTCOMES:
Leicester cough questionnaire | through study completion, average 1 year
  The LCQ is a validated 19-item cough-specific HRQoL questionnaire. It is divided into 3 domains (physical, social and psychological) and the overall score range from 3 to 21, with a higher score indicating a better cough related HRQOL.
The King's Brief Interstitial Lung Disease (KBILD) | through study completion, average 1 year
  The KBILD is a self-completed health status questionnaire that comprises of 15 items with the following three domains: psychological, breathlessness and activities and chest symptoms. Total score ranges from 0 to 100; 100 representing the best health status. This KBILD has an established minimal clinically important difference of 5-points in people with ILD.
Modified Borg scale (mBorg) | through study completion, average 1 year
  The modified Borg scale is widely used to assess the intensity of dyspnoea in individuals with chronic respiratory diseases and has recently been successfully adopted to assess the urge to cough and severity of cough in this population. The mBorg is measured on a 10 point scale; with 0 as feelings of "nothing at all" (no signs of dyspnoea) to 10 as "very very hard" intensity of dyspnoea.
Cough Hypersensitivity Questionnaire (CHQ) | through study completion, average 1 year
  The presence of triggers and laryngeal symptoms associated with cough were recorded using a standardized novel questionnaire, the CHQ. The CHQ comprises 23 items related to cough triggers, urge and laryngeal sensations associated with cough.
Functional Assessment of Chronic Illness Therapy Fatigue Scale (FACIT-F) | through study completion, average 1 year
  The FACIT-F is, a multi-dimensional 13-item questionnaire assessing tiredness, weakness and difficulty in handling daily living activities due to fatigue, over the previous 7 days. Participants are asked to rate their level of fatigue on a 4-point scale, where 0-not very much to 4- very much so. The sum of these values will provide a FACIT-F score ranging 0 to 52 (less fatigue to most fatigue).
Global rating of change questionnaire (GRCQ) | through study completion, average 1 year
  The GRCQ is a 15-point scale widely used to determine the participants' and health. professionals' perceptions about cough changes after interventions. Participants will be asked to rate global changes in cough in a scale ranging from -7 (a great deal worse) to +7 (a great deal better).
Satisfaction of cough therapy program | through study completion, average 1 year
  Participants' satisfaction and perceived benefits will be evaluated following completion of the intervention participants with a 9-item survey previously used to assess interventions in chronic respiratory diseases. The survey asks participants to report their level of agreement with statements on enjoyment and perceived improvements/benefits according to a 5-point Likert type scale (1=strongly agree; 5=strongly disagree).

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - West Park Healthcare Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chamberlain Mitchell SA, Garrod R, Clark L, Douiri A, Parker SM, Ellis J, Fowler SJ, Ludlow S, Hull JH, Chung KF, Lee KK, Bellas H, Pandyan A, Birring SS. Physiotherapy, and speech and language therapy intervention for patients with refractory chronic cough: a multicentre randomised control trial. Thorax. 2017 Feb;72(2):129-136. doi: 10.1136/thoraxjnl-2016-208843. Epub 2016 Sep 28. PMID 27682331